CLINICAL TRIAL: NCT05573594
Title: Efficiency of Muscle Energy Techniques In Female Patients Mechanical Lower Pain: A Randomised Control Trial A Randomised Control Trial
Brief Title: Efficiency of Muscle Energy Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sanem ŞENER, Principal Investigator, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIR
Record Dates: First submitted 2022-10-05; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Mechanical Low Back Pain
Keywords: Efficiency; Mechanical Low Back Pain; Muscle Energy Techniques
MeSH Terms: conditions — Low Back Pain | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MET Group (Experimental): the participants in the study group were under 8 sessions of MET, 2 times a week, in addition to the conventional physiotherapy program.
  In the content of conventional physiotherapy program for both groups; Hot Pack (20 min), Ultrasound (ITO brand 1 MHz and 1.5 W/cm2, 5 min), Transcutaneous Electrical Nerve Stimulation (TENS, 50-100 Hz, 20 min) and standard home exercises were included. The program went 5 times a week, 10 consecutive sessions. Each session lasted an average of 45 minutes.
  Interventions: Other: Muscle Energy Technique; Other: conventional physical therapy and rehabilitation
- Control Group (Experimental): In this study, the participants in the control group were under conventional physiotherapy program for 5 times a week, a total of 10 sessions
  In the content of conventional physiotherapy program for both groups; Hot Pack (20 min), Ultrasound (ITO brand 1 MHz and 1.5 W/cm2, 5 min), Transcutaneous Electrical Nerve Stimulation (TENS, 50-100 Hz, 20 min) and standard home exercises were included. The program went 5 times a week, 10 consecutive sessions. Each session lasted an average of 45 minutes
  Interventions: Other: conventional physical therapy and rehabilitation

INTERVENTIONS:
Other: Muscle Energy Technique — The Janda method (Post isometric relaxation PIR Technique), one of the Muscle Energy Techniques, was used on m.piriformis, m.quadratus lumborum, m.hamstring, m.psoas major muscles in the study group. First, the dysfunctional muscle was stretched passively by the physiotherapist up to the movement barrier, and 5-7 seconds of isometric muscle contraction in the opposite direction was requested from the patient at the barrier. This practice was continued until muscle tension or joint dysfunction disappeared.
  All participants performed standard home exercises consisting of stretching and strengthening. These exercises were taught to the participants by the physiotherapist in the first treatment session, and when they came to each treatment session, it was questioned whether they did it or not, and a control chart was created for exercise follow-up.
  Arms: MET Group
Other: conventional physical therapy and rehabilitation — In the content of conventional physiotherapy program for both groups; Hot Pack (20 min), Ultrasound (ITO brand 1 MHz and 1.5 W/cm2, 5 min), Transcutaneous Electrical Nerve Stimulation (TENS, 50-100 Hz, 20 min) and standard home exercises were included. The program went 5 times a week, 10 consecutive sessions. Each session lasted an average of 45 minutes.

SUMMARY:
Purpose: The aim of this study is to investigate the efficiency of the Muscle Energy Technique in female patients with mechanical low back pain.

Methods: A total of 40 female participants aged 30-45 were randomly divided into two groups (Study Group and Control Group). Control group participants were under 10 sessions conventional physical therapy and rehabilitation (TENS, US, hot pack) and performed standard home exercises. Study Group participants were under 8 sessions muscle energy technique in addition to conventional physical therapy and standard home exercises. Pain (Visual Analog Scale-VAS), spinal mobility (Modify Schober Test-MST), flexibility (Fingertip Floor Distance-FFD, Right and Left Lateral Flexion Floor Distance-LFFD), quality of life (Nottingham Health Profile-NHP), disability (Oswestry Disability Index-ODI), kinesiofobia (Tampa Kinesiofobia Scale-TKS) and depressive symptoms (Beck Depression Inventory-BDI) were measured at baseline, after the treatment and 3th months.

DETAILED DESCRIPTION:
There are many epidemiological and statistical studies showing the high incidence and prevalence of low back pain, which is a common problem all over the world (Manga et al 1993). Mechanical causes constitute 90% of the factors that cause low back pain (Diamond and Borenstein 2006).

Mechanical Low Back Pain (MLBP) is musculoskeletal pain of soft tissue origin that can be seen in the posterior lumbal region, sacral region or paraspinal region. MLBP, which is characterized by tendonitis, trigger points and muscle spasms, increases with movement and decreases with rest.

Muscle Energy Technique (MET) is a manual therapeutic procedure that creates voluntary contractions in skeletal muscles by creating force against the practitioner by the patient. MET is used to lengthen shortened muscles, mobilize restricted joints, and strengthen physiologically weakened muscles (Chaitow 2013).

Treatment methods generally applied to patients diagnosed with MLBP; physical therapy modalities, manual techniques, exercise therapy, medical therapy, psychological therapy and patient education. It is recommended that MET be used to reduce pain when administered to the spine (Wilson 2003) or muscles (Ballantyne et al. 2003).

The aim of our study is to investigate the efficiency of Muscle Energy Technique on spinal mobility, flexibility, pain, disability, fear avoidance behavior, quality of life and depressive symptoms in female patients with mechanical low back pain.

ELIGIBILITY:
Inclusion Criteria:

* being a volunteer female between the ages of 30 and 45
* having a complaint of low back pain for at least 3 months with the diagnosis of mechanical low back pain

Exclusion Criteria:

* having previous spinal surgery
* having radicular type low back pain
* having neuromuscular disease

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 8 week
  The pain severity felt by the participants in the lumbal region was evaluated with the Visual Analog Scale (VAS). VAS is the most appropriate tool for defining pain severity or intensity with its simplicity, reliability and validity as well as ratio scale features (Yakut and Kayıhan 2002). The VAS is a 10cm horizontal scale with 0 as "no pain" and 10 "very severe pain". The participant was asked to mark the severity of low back pain on the line. The marked point was measured and recorded.
Modified Shober Test | 8 week
  The participant's sacrum bases were combined with a line, the central point of this line was marked, 10 cm above and 5 cm below the central line were marked, and the participants were asked to bend fully forward without bending their knees. If the difference in this distance is less than 5 cm, the measurement was accepted as a decrease in spinal mobility (Tousignant 2005).
Fingertip-Ground Distance | 8 week
  In this test, the participant measures 15 cm. height, while standing upright on a block, he was asked to bend forward without bending his knees, and the fingertip-to-floor distance was measured with a tape measure (İnanoğlu and Baltacı 2014).
Lumbal Lateral Flexion Distance | 8 week
  It was started with the participant's feet shoulder-width apart, while standing upright, arms parallel to each other and at the side of the trunk. The place of the distal end of the middle finger of the right and left hand of the participant on the thigh was marked, and he was asked to tilt his body to the side by sliding his hand down on the thigh. The end point was marked again and the distance between the Right and Left LuMLBPr Lateral Flexion Distance and the ground was measured with a tape measure and the value found was recorded in centimeters (İnanoğlu and Baltacı 2014).
Tampa Kinesiophobia Scale | 8 week
  It was used to evaluate the fear avoidance levels (kinesiophobia) of the participants. This scale, which is used in acute and chronic low back pain, fibromyalgia and musculoskeletal injuries and whiplash-related diseases, consists of 17 questions and a 4-point Likert score (1 = strongly disagree, 4 = completely agree) is used. Items 4, 8, 12, and 16 are reverse-scored, and the high score of the participant in the scale, which is calculated with a total score of 17-68, indicates that kinesiophobia is also high (Yılmaz 2011).
Oswestry Disability Index | 8 week
  It was used to evaluate the disability level. The Turkish validity and reliability of this index was done by Yakut et al. (Yakut 2004). In the anMET, which questions the disability status in activities of daily living (pain severity, personal care, lifting, walking, sitting, standing, sleeping, social life, travel, and the degree of change in pain), with an index consisting of 10 items, those who score 0-14 score mild, 15- Those with a score of 29 were considered to have moderate disability, and those with a score above 30 were considered to have advanced disability (Fairbank 2000).
Nottingham Health Profile | 8 week
  The Turkish version of Küçükdeveci et al. was used to evaluate the health-related quality of life of the participants and to measure the extent to which the health problems perceived by the individual affect normal daily activities. In the questionnaire, which evaluates health status in 6 dimensions with 38 items, energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items) and consists of physical activity (8 items). When the scores obtained from the sub-scores for the total NSP score approach from 0 to 100, it is accepted that the quality of life decreases (Küçükdeveci 2000).
Beck Depression Inventory | 8 week
  This questionnaire, the Turkish validity and reliability of which was conducted by Hisli et al. in 1988, was used to evaluate the depressive symptoms of the participants. Somatic, cognitive, motivational and emotional symptoms are scored with a total of 21 items. An increase in the total scores of the participants indicates an increase in their depressive symptoms (Beck et al. 1961). In our study, analysis was performed using the total scores of the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diamond S, Borenstein D. Chronic low back pain in a working-age adult. Best Pract Res Clin Rheumatol. 2006 Aug;20(4):707-20. doi: 10.1016/j.berh.2006.04.002. PMID 16979534
- [Background] Fryer G, Pearce AJ. The effect of muscle energy technique on corticospinal and spinal reflex excitability in asymptomatic participants. J Bodyw Mov Ther. 2013 Oct;17(4):440-7. doi: 10.1016/j.jbmt.2013.05.006. Epub 2013 May 30. PMID 24139001